CLINICAL TRIAL: NCT00522340
Title: Anti-Arrhythmic Effects of Exercise After an Implantable Cardioverter Defibrillator (ICD)
Brief Title: Exercise After an ICD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Cindy Dougherty, Professor, Biobehavioral Nursing and Health Systems, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31202-B; R01HL084550-01A1 (NIH)
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Defibrillators, Implantable; Heart Failure, Congestive
Keywords: Implantable Cardioverter Defibrillators; ICD; Exercise; Cardiac; Inflammation
MeSH Terms: conditions — Heart Failure; Motor Activity; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobic Exercise Program (Experimental)
  Interventions: Behavioral: Aerobic Exercise Program
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Aerobic Exercise Program — Home walking 1 hour a day for 5 days/week for 8 weeks. Then 30 minutes a day on all or most days of the week.
  Arms: Aerobic Exercise Program

SUMMARY:
An implantable cardioverter-defibrillator (ICD) is a small device that is surgically implanted in the chest or abdomen and uses electrical pulses or shocks to help control life-threatening, irregular heartbeats. Increasing aerobic exercise may provide health benefits to people with ICDs. This study will examine the effects of an exercise program on heart and lung function in people who have an ICD.

DETAILED DESCRIPTION:
An ICD is a device designed to quickly detect a life-threatening, rapid heartbeat. Through a process called defibrillation, the ICD tries to convert an abnormal heart rhythm back to normal by delivering an electrical shock to the heart. The ICD continuously monitors heartbeats to ensure that they are normal, and it only delivers a shock to the heart when it senses a life-threatening rhythm. People who have experienced ventricular fibrillation, which is a severely abnormal heart rhythm, or ventricular tachycardia, which is a rapid heart beat that begins in the bottom chambers of the heart, are common recipients of an ICD. Other potential ICD recipients include people who have survived a heart attack, but have weak hearts; people with heart muscle problems; and people with reduced pumping function in their heart. People who have ICDs may benefit from aerobic exercise to improve their physical fitness and overall health. The purpose of this study is to evaluate the effectiveness of an exercise program at improving heart and lung function in people who have an ICD.

In this 6-month study, participants will be randomly assigned to either take part in the exercise program or receive usual care. At a baseline study visit, all participants will complete an exercise treadmill test, wear a Holter monitor to record heart activity for 24 hours, undergo blood collection, and complete questionnaires to assess quality of life, anxiety, and depression. Participants taking part in the exercise program will receive 1 hour of exercise education over the telephone. During Weeks 1 through 8, participants will stretch for 10 minutes and walk 1 hour daily for 5 days a week; during Weeks 9 through 24, participants will walk 30 minutes daily for 5 days a week. Participants will wear a Polar Heart Rate monitor to record their heart rate and a pedometer to keep track of the number of steps walked. They will also record details of their exercise in a daily activity log. Throughout the entire study, a study nurse will call participants on a weekly basis to check on their progress and to help resolve any exercise-related problems. At Weeks 8 and 24, all participants including those receiving usual care, will attend a study visit for repeat baseline evaluations. Study researchers will review medical records to collect various information, including the reason for needing an ICD, the type and settings of the ICD, medication use, medical history, current health problems, lab test results, echocardiogram images of the heart, and electrocardiogram (EKG) results.

ELIGIBILITY:
Inclusion Criteria:

* ICD implanted in the 12 months prior to study entry
* Currently taking beta blocker medication
* Speaks and reads English

Exclusion Criteria:

* Unstable angina, heart attack, or percutaneous coronary intervention (PCI) in the 3 months prior to study entry
* Experienced an ICD shock in the 3 months prior to study entry
* Currently exercises 3 times a week for 20 minutes a day
* Alcohol Use Disorders Identification Test-Consumption (AUDIT-C) score for alcohol consumption greater than 4
* Shore Blessed score for cognitive dysfunction greater than 6

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2007-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary function | Measured at Week 8

SECONDARY OUTCOMES:
Heart rate variability | Measured at Week 8
Quality of life | Measured at Weeks 8 and 24
Anxiety | Measured at Weeks 8 and 24
Depression | Measured at Weeks 8 and 24
Interleukin-6 (IL-6) | Measured at Weeks 8 and 24
B-type natriuretic peptide (BNP) | Measured at Weeks 8 and 24
ICD shocks | Measured at Weeks 8 and 24
Tissue necrosis factor-alpha (TNF-alpha) | Measured at Weeks 8 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Dougherty, ARNP, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Dougherty CM, Cordoza M, Wang D, Alsoyan AH, Stein PK, Burr RL. Aerobic Exercise Improves Heart Rate Variability After an Implantable Cardioverter Defibrillator (ICD). Biol Res Nurs. 2024 Oct;26(4):584-596. doi: 10.1177/10998004241261273. Epub 2024 Jun 16. PMID 38881252
- [Derived] Dougherty CM, Burr RL, Kudenchuk PJ, Glenny RW. Aerobic Exercise Effects on Quality of Life and Psychological Distress After an Implantable Cardioverter Defibrillator. J Cardiopulm Rehabil Prev. 2020 Mar;40(2):94-101. doi: 10.1097/HCR.0000000000000444. PMID 31397768
- [Derived] Dougherty CM, Luttrell MN, Burr RL, Kim M, Haskell WL. Adherence to an Aerobic Exercise Intervention after an Implantable Cardioverter Defibrillator (ICD). Pacing Clin Electrophysiol. 2016 Feb;39(2):128-39. doi: 10.1111/pace.12782. Epub 2015 Dec 3. PMID 26548341
- [Derived] Dougherty CM, Glenny RW, Burr RL, Flo GL, Kudenchuk PJ. Prospective randomized trial of moderately strenuous aerobic exercise after an implantable cardioverter defibrillator. Circulation. 2015 May 26;131(21):1835-42. doi: 10.1161/CIRCULATIONAHA.114.014444. Epub 2015 Mar 19. PMID 25792557
- [Derived] Nguyen HQ, Steele BG, Dougherty CM, Burr RL. Physical activity patterns of patients with cardiopulmonary illnesses. Arch Phys Med Rehabil. 2012 Dec;93(12):2360-6. doi: 10.1016/j.apmr.2012.06.022. Epub 2012 Jul 5. PMID 22772084